CLINICAL TRIAL: NCT06919796
Title: Systems Biology of a mRNA Vaccine Against Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Given Via Intradermal (ID) Injection Using Tropis Needle-Free Injection System (NFIS) or Intramuscular (IM) Injection Using Needle and Syringe
Brief Title: mRNA Covid-19 Vaccine Immune Response Comparisons Using Different Delivery Routes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaJet, Inc. (Industry)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVID-PJ-01
Record Dates: First submitted 2025-04-03; First posted 2025-04-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Evaluate Immune Responses Following mRNA COVID-19 Vaccine Administration Through Different Delivery Routes in Healthy Volunteers; SARS CoV-2
Keywords: Tropis ID; Needle-free injection; Tropis
MeSH Terms: interventions — BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- mRNA vaccine administration via Tropis ID NFIS (Experimental): Immunization with a single dose of mRNA Covid-19 vaccine administered intradermally using the Tropis Needle Free Injection System
  Interventions: Biological: COMIRNATY®
- Intramuscular injection of the mRNA Covid-19 vaccine via needle and syringe (Active Comparator): Immunization with a single dose of mRNA Covid-19 vaccine administered intramuscularly using needle and syringe
  Interventions: Biological: COMIRNATY®

INTERVENTIONS:
Biological: COMIRNATY® — COVID-19 Vaccine, mRNA suspension

SUMMARY:
The purpose of this study is to determine if immune responses differ when the mRNA COVID-19 vaccine is given through different delivery methods, including a needle-free injection system, or via intramuscular injection using needle and syringe

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and give informed consent
2. Adults aged 18 to 50 years old.
3. Willing and able to comply with all scheduled visits, vaccination, and laboratory tests.
4. Determined by investigator to be in good health based on medical history, targeted physical exam and laboratory testing.
5. Participants with pre-existing stable chronic medical conditions defined as condition not requiring significant change in therapy or hospitalization for worsening disease within 4 weeks from enrollment, can be included at the discretion of the investigator.
6. For women of childbearing potential: willing to engage in effective methods of contraception starting at least 30 days prior to enrollment and for the duration of the study.

Exclusion Criteria:

1. Receipt of blood products 90 days prior to study entry and for the duration of the study.
2. Volunteers who donated blood 60 days before screening OR will donate blood on or before D30.
3. Receipt of any experimental agents within 30 days or 5 half-lives whichever is longer prior to vaccination and for the duration of the study.
4. Receipt of any licensed vaccine within 60 days prior to study vaccination or planned receipt of any vaccine until 60 days later as well as receipt of COVID-19 vaccine for the duration of the study.
5. Receipt of a COVID-19 vaccine or confirmed COVID-19 in the past year or positive SARS-CoV-2 antigen test on vaccination day.
6. Chronic medical problems including (but not limited to) autoimmune disease, severe gastrointestinal disease, and grade 4 hypertension.
7. Any diseases or conditions that put individuals at increased risk for severe COVID-19 illness, including: type 1 or 2 diabetes, chronic lung disease (including moderate to severe asthma, bronchiectasis, bronchopulmonary dysplasia, chronic obstructive pulmonary disease (COPD), interstitial lung disease including idiopathic pulmonary fibrosis, pulmonary embolism, or pulmonary hypertension), cystic fibrosis, dementia, Parkinson's disease, cerebrovascular disease, chronic liver disease, chronic kidney disease (any stage), heart conditions, hemoglobin blood disorders (sickle cell disease, thalassemia).
8. BMI > 40 kg/m2
9. Any potentially immune mediated disease (with the exception of well controlled hypothyroidism).
10. Alcohol or drug abuse and psychiatric conditions that in the opinion of the investigator would preclude compliance with the trial or interpretation of safety or endpoint data.
11. Impaired immune function or chronic infections including (but not limited to) HIV, hepatitis B or C; organ transplant; active cancer or any history of hematologic cancer; receipt of chemotherapy, radiation therapy (past 12 months) or any other potentially immunosuppressive therapy [i.e. received oral, intramuscular or intravenous systemic immunosuppressants, or immune modifying drugs for >14 days in total within 6 months prior to any study vaccine dose (for corticosteroids ≥ 20 mg/day of prednisone equivalent). Note: Topical medications are allowed.], congenital immunodeficiency, anatomical or functional asplenia.
12. Pregnancy or breast feeding or planned pregnancy for the duration of the study.
13. Severe reactions to prior vaccination with Covid-19 mRNA vaccine or any of its components, including anaphylaxis.
14. History of Guillain Barré syndrome or myopericarditis.
15. Volunteers with any acute illness, including any fever (> 100.4 F [> 38.0C], regardless of the route) within 3 days prior to study entry.
16. Social, occupational, or any other condition that in the opinion of the investigator might interfere with compliance with the study and vaccine evaluation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | Nine months
  In 40 participants response rate, and magnitude of SARS-CoV-2-specific antibody neutralization titers will be measured at Day 30 and Month 6-9 after vaccination

SECONDARY OUTCOMES:
Secondary Objective | Nine months
  1. Percentage of participants with solicited injection site and systemic AEs within 7 days after vaccination.
  2. Percentage of participants with unsolicited AEs until Day 30 after vaccination.
  3. Percentage of participants with SAEs, MAAEs and AEs leading to study withdrawal throughout the entire study period.
  4. Percentage of participants with AESIs (Appendix A) throughout the entire study period.
  5. Percentage of participants with grade 2 and above AEs within 7 days after each fine needle aspirates of draining lymph nodes and bone marrow aspirates.

CONTACTS AND LOCATIONS:
Locations (1):
- Hope Clinic of the Emory Vaccine Center Division of Infectious Diseases, Department of Medicine, School of Medicine, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Principal Investigator has confirmed IPD will not be shared with other reserchers